CLINICAL TRIAL: NCT07091877
Title: Cognitive Reappraisal for Mitigating Incubation of Cocaine Cue-Reactivity
Brief Title: Cocaine Cue-reactivity Incubation Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Muhammad Parvaz, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY-22-01618; R01DA058039 (NIH)
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-12

CONDITIONS: Cocaine Use Disorder
Keywords: Cocaine; Craving; EEG; Cue-reactivity; Cognitive reappraisal; Incubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Reappraisal (CR+) (Experimental): Participants in this arm will complete the Cognitive Reappraisal task repeatedly at 2 weeks, 1-2 months, 3 months, and 5 months after abstinence initiation.
  Interventions: Behavioral: Cognitive Reappraisal
- No Cognitive Reappraisal (CR-) (Sham Comparator): Participants in this arm will complete a control cue-reactivity task repeatedly at 2 weeks, 1-2 months, 3 months, and 5 months after abstinence initiation.
  Interventions: Behavioral: Control cue-reactivity task

INTERVENTIONS:
Behavioral: Cognitive Reappraisal — Cognitive Reappraisal (CR) is a cognitive-behavioral technique and will complete the Cognitive Reappraisal task.
  Arms: Cognitive Reappraisal (CR+)
Behavioral: Control cue-reactivity task — Participants will complete a control cue-reactivity task.
  Arms: No Cognitive Reappraisal (CR-)

SUMMARY:
In this study, the research team proposes to longitudinally assess incubation of cue-reactivity, its reduction with cognitive reappraisal (CR; a self-regulation technique) and examine the impact of CR on clinical outcomes in individuals with cocaine use disorder (CUD). The primary objective is to use psychophysiological markers for tracking brain activity and behavior and changes therein with the use of CR during abstinence in CUD. The secondary objective is to examine whether brain and behavioral changes are associated with clinical outcomes in individuals with CUD. The primary endpoint is the time-related change in brain and behavioral indices with CR during abstinence in individuals with CUD. The secondary endpoint is the impact of CR-mediated changes on clinical outcomes of individuals with CUD.

In this 5-yearlong study the research team will recruit 252 individuals seeking-treatment for CUD, 126 of whom will be randomly assigned to complete the Cognitive Reappraisal task repeatedly at 2 weeks, 1-2 months, 3 months, and 5 months after abstinence initiation (CR+ group), and the other 126 will be assigned to complete a Control task at the same time points (CR- group). All individuals between the ages of 18 and 65 years, irrespective of sex and sexual orientation will be recruited. Participation in the research study will be 5 sessions taking place (one at 2 weeks from screening, one at a month from screening, one at 3 months from screening, one at 5 months from screening, and one the month after the 5 month session) over the course of 6 months.

The study will include EEG testing and will be administered multiple times over the course of 6 months. Participants will be randomized to one of the two groups; one group will get the Cognitive Reappraisal (CR+) intervention and the other group will get a Control intervention (CR-).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and give informed consent
* Age 18-65
* DSM-5 Diagnosis of CUD (Cocaine Use Disorder)
* Have appropriate abstinence duration (i.e., <2 months) at the first visit.
* Must be seeking treatment for CUD (at the first visit)

Exclusion Criteria:

* DSM-5 diagnosis for other psychiatric illnesses (other than mood and anxiety disorders that are highly comorbid with substance use disorders)
* Urine positive for any psychoactive drugs (e.g., cocaine, methamphetamine, cannabis, opiates, benzodiazepines, etc.) at baseline
* Head trauma with loss of consciousness
* History of neurological diseases, including seizures
* Thick and/or non-removable hair braids that present difficulty for EEG electrode-scalp contact

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Late Positive Potential (LPP) amplitude | <2 months, 3 months, and 5 months after abstinence initiation
  EEG-derived Late Positive Potential (LPP) amplitude will be measured while participants view cocaine-related cues. Higher amplitudes indicate greater cue reactivity.

SECONDARY OUTCOMES:
Change in Late Positive Potential (LPP) amplitude with CR | <2 months, 3 months, and 5 months after abstinence initiation
  EEG-derived Late Positive Potential (LPP) amplitude changes during cocaine cue exposure while using cognitive reappraisal techniques.
Changes in cocaine abstinence duration | <2 months, 3 months, and 5 months after abstinence initiation
  Cocaine abstinence (measured in number of days) will be assessed via Timeline Followback Calendar, which tabulates the number of days cocaine was used in the past 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad A Parvaz, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Anyone who wishes to access the data. For individual participant data meta-analysis. Data are available indefinitely at URL below.
URL: https://openneuro.org/